CLINICAL TRIAL: NCT03073811
Title: Nutritional (High Protein) Perihabilitation in Older Veterans Undergoing Surgery
Brief Title: Nutritional Perihabilitation in Older Veterans Undergoing Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: E2348-W; IK2RX002348 (NIH)
Record Dates: First submitted 2017-02-23; First posted 2017-03-08 (Actual); Results first posted 2024-01-31 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Malnutrition; Nutritional Risk; Abdominal Surgery
Keywords: protein supplementation; older adults; nutrition perihabilitation; perioperative optimization; Veterans
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PeriHab (Experimental): Provided nutrition counseling and prescribed to consume 1.6 g/kg/body weight as well as provided 30 grams of high quality protein three times per day for two weeks before and four weeks after surgery.
  Interventions: Dietary Supplement: Protein enhanced nutrition intervention
- PoshControl (Active Comparator): Provided nutrition counseling and prescribed to consume 1.0 g/kg/body weight in the form of educational handouts explained by a Registered Dietitian and one oral nutrition supplement per day for two weeks before surgery.
  Interventions: Other: Education Control

INTERVENTIONS:
Dietary Supplement: Protein enhanced nutrition intervention — Participants will be provided 30 grams of high quality protein (Ensure Max) three times a day for two weeks before surgery and four weeks after surgery.
  Other Names: Perihabilitation
  Arms: PeriHab
Other: Education Control — provided educational on the role of nutrition to prepare for and heal from surgery, and Registered Dietitian will instruct participant to follow instruction on handout and one oral nutrition supplement per day for two week before surgery.
  Other Names: PoshControl
  Arms: PoshControl

SUMMARY:
This research study will be conducted in two parts. The first part will consist of selecting appropriate screening and assessment tools for Veterans undergoing elective surgery and identifying the number of Veterans who are malnourished and at risk of malnutrition. The second portion of the study will be to determine if a protein-enhanced diet before and after surgery will improve function and postoperative outcomes and compare the results to an education control group.

DETAILED DESCRIPTION:
In year 1 of the two-part research study, an observational, prospective study of 75 Veterans preparing for elective surgery will be conducted. The purpose of this study will be to select appropriate nutrition screening and assessment tools and to employ them to characterize malnutrition prevalence and severity and establish cut-off values associated with malnutrition in this population. In years 2-5 of the research two-part research study, a pilot randomized controlled trial will be conducted. The purpose of this study will be evaluate the feasibility, fidelity, and acceptability of a perioperative protein-enhanced intervention compared to an educational control. Veterans who are malnourished or at risk of being malnourished will be randomly assigned on a 1:1 ratio to either an education (nutritional counseling) control or high-protein perihabilitation arm. Participants in the high-protein perihabilitation arm will be provided with 30 grams of high quality protein supplements three times per day. The study will take place two weeks prior to an elective abdominal or GI surgery and will continue 4 weeks post surgery.

ELIGIBILITY:
Inclusion Criteria:

* Elective abdominal surgery

  * upper GI
  * colorectal
  * hepatobiliary
  * pancreatic
  * intra-abdominal
  * Abdominal aortic aneurysm
* Referred to the VA Perioperative Optimization of Senior Health Clinic
* Able to record dietary intake or has a proxy who can record dietary intake

Exclusion Criteria:

* Cognitive impairment
* Unwillingness to be randomized to either intervention arm, submit to study testing, or continuously participate in the intervention for six weeks
* Living in skilled nursing facility
* No access to telephone

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn N. Starr, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- PeriHab: Provided nutrition counseling and prescribed to consume 1.6 g/kg/body weight as well as provided 30 grams of high quality protein three times per day for two weeks before and four weeks after surgery.
  Protein enhanced nutrition intervention: Participants will be provided 30 grams of high quality protein three times a day for two weeks before surgery and four weeks after surgery.
Period: Overall Study
Arm/Group | PeriHab | PoshControl
Started | 26 | 24
Completed | 19 | 16
Not Completed | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PeriHab | PoshControl | Total
Number analyzed (Participants) | 26 | 24 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.8 (6.6) | 73.9 (5.9) | 73.9 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 24 | 24 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 5 | 19
  White | 12 | 19 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26 | 24 | 50
Short Physical Performance Battery [Mean (Standard Deviation); unit: units on a scale] — SPPB total score is on a scale from 0 to 12, with a higher score indicating better physical function.
  units on a scale | 8.2 (2.6) | 7.9 (2.4) | 8.1 (2.5)
Cancer Diagnosis [Count of Participants; unit: Participants] | 16 | 15 | 31
Body weight, lbs [Mean (Standard Deviation); unit: lbs] | 177.4 (32.9) | 195.1 (48.6) | 189.9 (41.7)
Body Mass Index, kg/m^2 [Mean (Standard Deviation); unit: kg/m2] | 26.4 (4.1) | 28.5 (6.6) | 27.4 (5.5)

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Feasibility of a Perioperative Protein-enhanced Intervention Compared to Control Arm.
Description: Feasibility was measured as retention. Hypothesis was that 80% of the participants would be retained.
Time Frame: day of surgery (an average of 12 days from baseline [midpoint]) and 30-day post-surgery (endpoint)
Measure: Count of Participants; unit: Participants
Arm/Group | PeriHab | PoshControl
Number analyzed (Participants) | 26 | 24
Participants
  Day of Surgery | 23 | 20
  Postoperative Follow-up | 19 | 16

2. Primary Outcome: Determine Acceptability of Perioperative Protein-enhanced Intervention Compared to an Educational Control
Description: Satisfaction of overall participation in the research study (Likert Scale). I am glad I participated in this research study. 1 - Strongly Disagree and 5- Strongly Agree
Time Frame: 30-day post-surgery follow-up (endpoint)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PeriHab | PoshControl
Number analyzed (Participants) | 19 | 16
units on a scale | 4.6 (0.6) | 4.9 (0.3)

3. Primary Outcome: Physical Function
Description: Short physical performance battery - higher scores means a better physical performance (Total score = 0-12)
Time Frame: Baseline, day of surgery (an average of 12 days from baseline), 30-days post-surgery
Population: Perihab (midpoint; n=23) - surgery was cancelled (n=3) PoshControl (midpoint; n=18) - surgery was cancelled (n=3), dropped (n=1); surgery time changed (n=2) Perihab (endpoint; n=18) - surgery was cancelled morning of surgery (n=2); death (n=1); COVID (n=2) PoshControl (n=16; endpoint) - surgery was cancelled morning of surgery (n=2); death (n=1); hospitalization (n=1)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PeriHab | PoshControl
Number analyzed (Participants) | 26 | 24
score on a scale
  Baseline | 8.2 (2.6) | 7.9 (2.4)
  Morning of Surgery (midpoint): number analyzed (Participants) | 23 | 18
  Morning of Surgery (midpoint) | 9.7 (2.3) | 9.0 (2.0)
  30 day postop (endpoint): number analyzed (Participants) | 18 | 16
  30 day postop (endpoint) | 9.0 (2.9) | 8.8 (2.3)

4. Secondary Outcome: Hospital Readmission
Description: determine from medical records
Time Frame: endpoint (30 days post-surgery)
Reporting Status: Not Posted, anticipated posting 2025-06

5. Secondary Outcome: Dietary Intake
Description: Three day food records will be collected.
Time Frame: baseline, day of surgery (midpoint), 30-day post-surgery (endpoint)
Reporting Status: Not Posted, anticipated posting 2025-06

6. Secondary Outcome: Handgrip Strength
Description: Hand dynamometer will be used to determine grip strength. Maximum grip strength will be determined by conducting two trials on the dominant hand, with 30 second rest between trials.
Time Frame: baseline, day of surgery (midpoint), 30-day post-surgery (endpoint)
Reporting Status: Not Posted, anticipated posting 2025-06

7. Secondary Outcome: Nutritional Risk Screener-2002
Description: Validated Nutritional Risk Screener-2002 Questionnaire to determine nutritional risk
Time Frame: baseline, day of surgery (midpoint), 30-day post-surgery (endpoint)
Reporting Status: Not Posted, anticipated posting 2025-06

8. Secondary Outcome: Patient Generated-Subjective Global Assessment
Description: Validated Patient Generate Subjective Global Assessment Questionnaire to determine malnutrition status
Time Frame: baseline, day of surgery (midpoint), 30-day post-surgery (endpoint)
Reporting Status: Not Posted, anticipated posting 2025-06

9. Secondary Outcome: Discharge Location
Description: determine from medical records
Time Frame: endpoint (30 days post-surgery)
Reporting Status: Not Posted, anticipated posting 2025-06

10. Secondary Outcome: Length of Stay
Description: determine from medical records
Time Frame: endpoint (30 days post-surgery)
Reporting Status: Not Posted, anticipated posting 2025-06

11. Secondary Outcome: Emergency Department Readmission
Description: Prevalence of emergency department admissions following surgery.
Time Frame: endpoint (30 days post-surgery)
Reporting Status: Not Posted, anticipated posting 2025-06

12. Secondary Outcome: Postoperative Complications
Description: determine from medical records
Time Frame: endpoint (30 days post-surgery)
Reporting Status: Not Posted, anticipated posting 2025-06

13. Secondary Outcome: Albumin, g/dL
Description: A measure of protein in the blood. Lower level may indicate infection or inflammation.
Time Frame: baseline, day of surgery (midpoint), 30-day post-surgery (endpoint)
Reporting Status: Not Posted, anticipated posting 2025-06

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for each participant from enrollment to study completion or study withdraw. The duration of participation in the study was approximately 8 weeks.
Arm/Group | PeriHab | PoshControl
All-Cause Mortality (participants affected / at risk) | 1/26 | 1/24
Serious Adverse Events (participants affected / at risk) | 2/26 | 1/24
Other Adverse Events (participants affected / at risk) | 1/26 | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PeriHab (N=26) | PoshControl (N=24)
Surgery site infection (Surgical and medical procedures) | 1 (1) | 0 (0)
Shortness of Breath and Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PeriHab (N=26) | PoshControl (N=24)
Swelling in foot (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-13): https://cdn.clinicaltrials.gov/large-docs/11/NCT03073811/Prot_SAP_000.pdf